CLINICAL TRIAL: NCT06387199
Title: Alleviating Carbohydrate Counting Using Weekly Subcutaneous Semaglutide Injections in People with Type 1 Diabetes on Closed-Loop Insulin Therapy: a 2x4 Factorial Randomized Placebo-Controlled Trial
Brief Title: Alleviating Carbohydrate Counting for Patients with Type-1 Diabetes Using a Closed Loop System with Weekly Subcutaneous Semaglutide
Acronym: SEMA SMA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Assistant Professor, Endocrinology & Metaolism, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-10227
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus
Keywords: insulin; Closed-loop system; GLP-1 receptor agonist; Semaglutide; Diabetes mellitus, type 1; ozempic
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: randomized placebo-controlled crossover 2x3 factorial designed trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly placebo injections on regular closed-loop insulin pump therapy (Active Comparator)
  Interventions: Drug: Placebo with 4 meal strategies
- Weekly semaglutide (Ozempic®) injections on regular closed-loop insulin pump therapy (Experimental): Semaglutide is a Glucagon-like peptide 1 (GLP-1) receptor agonist. It up regulates GLP-1, which reduces glucagon levels, increases satiety and - in some particular cases - increases insulin production. It will be subcutaneously injected weekly by participants at progressively increasing doses. Once the maximum tolerated dose is achieved, participants will begin the meal strategies.
  Interventions: Drug: Semaglutide with 4 meal strategies

INTERVENTIONS:
Drug: Semaglutide with 4 meal strategies — The blinded drug will be used in addition to the participants routine closed-loop insulin pump therapy. It will be administered through subcutaneous injection on a weekly basis. The first 12 weeks will include progressively increasing doses of the drug whereby, the dose increases every 4 weeks. Once the maximum tolerated dose is achieved after 12 weeks, participants will undergo 4 meal strategies in a randomized order. These include (in no particular order); full carbohydrate counting with rapid-acting insulin, SMA with rapid-acting insulin, SMA with Lyumjev and fully closed-loop system with Lyumjev. Each meal strategy will be 3 weeks in duration and will occur sequentially in the designated order.
  Arms: Weekly semaglutide (Ozempic®) injections on regular closed-loop insulin pump therapy
Drug: Placebo with 4 meal strategies — The blinded drug will be used in addition to the participants routine closed-loop insulin pump therapy. It will be administered through subcutaneous injection on a weekly basis. The first 12 weeks will include progressively increasing doses of the drug whereby, the dose increases every 4 weeks. Once the maximum tolerated dose is achieved after 12 weeks, participants will undergo 4 meal strategies in a randomized order. These include (in no particular order); full carbohydrate counting with rapid-acting insulin, SMA with rapid-acting insulin, SMA with Lyumjev and fully closed-loop system with Lyumjev. Each meal strategy will be 3 weeks in duration and will occur sequentially in the designated order.
  Arms: Weekly placebo injections on regular closed-loop insulin pump therapy

SUMMARY:
A closed-loop insulin system, often labelled the "artificial pancreas" (AP), consists of an insulin pump, a continuous glucose monitor, and an interface coordinating between them to regulate insulin dosage based on glucose levels. Primarily designed for managing type 1 diabetes, this system has demonstrated significant benefits in previous studies. Yet, despite these advantages, certain challenges persist.

Semaglutide, utilized in treating type 2 diabetes and obesity, is a once-weekly injectable medication that elevates levels of a gastrointestinal hormone known as Glucagon-Like Peptide-1 (GLP-1). This hormone alters gastric emptying, inhibits glucagon release, and reduces appetite. While not officially sanctioned for type 1 diabetes treatment in North America, studies have explored its efficacy as an adjunctive therapy alongside insulin, yielding favorable outcomes in blood glucose regulation. Comparable drugs like liraglutide and exenatide have been employed in type 1 diabetes treatment as well, albeit with less pronounced glucose-regulating effects compared to semaglutide, even in type 2 diabetes.

The goal of this 50-week randomized placebo-controlled crossover 2x4 factorial designed trial is to assess whether commercial automated insulin delivery (AID) systems using rapid-acting insulin with adjunct weekly injections of semaglutide (at the maximally tolerated dose) can replace carbohydrate counting with simple meal announcements (SMA) without degrading glucose control.

DETAILED DESCRIPTION:
The main questions this study aims to answer are:

* Can weekly injections of semaglutide at the maximum tolerated dose in individuals with T1D on closed-loop therapy with SMA and rapid-acting insulin result in a non-inferior time spent in target range (3.9-10 mmol/L) compared to weekly placebo injections on closed-loop system with full carbohydrate counting.
* Can weekly injections of semaglutide at the maximum tolerated dose, in combination with ultra-rapid actin insulin (Lyumjev);

  1. Eliminate carbohydrate counting and any meal announcement (i.e fully closed-loop) in people with T1D on closed-loop therapy without degrading glucose control.
  2. Be more effective in substituting carbohydrate counting with SMA in people with T1D on closed-loop therapy compared with traditional rapid-acting insulin.

Participants will be asked to undergo two subsequent blinded drug interventions; one with semaglutide and the other with placebo. Both interventions include 4 meal strategies each with a 3-week duration; full carbohydrate counting with rapid-acting insulin, SMA with rapid-acting insulin, SMA with Lyumjev and fully closed-loop system with Lyumjev.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. A clinical diagnosis of T1D for at least one year, as per their treating diabetes physician in agreement with the primary investigator's clinical judgment (confirmatory C-peptide and antibodies will not be required)
3. Minimum 3-month use of a commercial advanced automated insulin delivery system. 4.4. Agreement to use an effective method of birth control for individuals with child-bearing potential. Child-bearing potential refers to participants of the female sex post-menarche who have not reached menopause and who do not have a medical condition causing sterility (e.g., hysterectomy). Post-menopausal state refers to the absence of menses for 12 months without any alternative cause.

Exclusion Criteria:

1. Use of GLP1-RAs within the last 4 weeks.
2. Use of any anti-hyperglycemic agent other than insulin within the last 2 weeks.
3. Planned or ongoing pregnancy
4. Breastfeeding
5. Severe hypoglycemic episode within the last 3 months, defined as an event where glucose was < 4 mmol/L resulting in seizure, loss of consciousness, or need to present to the emergency department
6. Severe diabetic ketoacidosis (DKA) within the last 6 months ("severe" referring to need to present to medical attention and requirement of intravenous insulin)
7. Prior history of acute pancreatitis, chronic pancreatitis, or gallbladder disease
8. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2
9. Severe impairment of renal function with eGFR <30 mL/min/1.73 m2 (using CKD-EPI formula), measured within the last 12 months
10. Clinically significant diabetic retinopathy or gastroparesis, as per the clinical judgment of the investigator
11. Bariatric surgery within the last 6 months.
12. A serious medical or psychiatric illness that is likely to interfere with study participation as per the judgment of the investigator (e.g. cirrhosis, active cancer, decompensated schizophrenia).
13. Body mass index ≤ 21 kg/m2
14. Inability or unwillingness to comply to safe diabetes management in the view of the study group (e.g. inappropriate treatment of hypoglycemia or lack thereof)
15. Concern for safety of the participant, as per the clinical judgment of the primary investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of daytime plasma glucose levels spent in target range (semaglutide vs. placebo) | 24 weeks
  Target range is defined to be between 3.9 and 10.0 mmol/L of plasma glucose for placebo vs semaglutide (at maximal tolerated dose) on closed-loop insulin therapy

SECONDARY OUTCOMES:
Percentage of time spent in the range of glucose levels between 3.9 and 7.8 mmol/L | 24 weeks
  % as per CGM data
Percentage of time spent in glucose levels below 3.9 and 3.0 mmol/L | 24 weeks
  % as per CGM data
Percentage of time spent in glucose levels above 7.8, 10 and 13.9 mmol/L | 24 weeks
  % as per CGM data
Mean glucose level | 24 weeks
  Defined as per CGM data, in mmol/L
Standard deviation of glucose levels as a measure of glucose variability | 24 weeks
  Defined as per CGM data, in mmol/L
Percentage coefficient of variation of glucose levels | 24 weeks
  % as per CGM data
Proportions of participants with time in range between 3.9 - 10.0 mmol/L≥ 70% | 24 weeks
  As per CGM data
Glycated hemoglobin (HbA1c) | 24 weeks
  Blood test to assess glucose control within 3-4 months
Area under the curve 0-2h post meal, 0-3h post peal | 24 weeks
  As per CGM data
Average scores between interventions on the Type 1 Diabetes Distress Scale questionnaire | 24 weeks
  17-item questionnaire with a 6-point Likert scale from 1 (no stress) to 6 (high stress) for each item. Total score obtained from summing the scores of all items
Average scores between interventions on the Diabetes Treatment Satisfaction questionnaire | 24 weeks
  8-item questionnaire with a 7-point Likert scale ranging from 0 (low satisfaction) to 6 (high satisfaction). Total score obtained from summing the scores of all items.
Average scores between interventions based on the Hypoglycemic Fear Survey - II | 24 weeks
  33-item questionnaire with a 5-point Likert scale ranging from 1 (never) to 5 (almost always). Total score obtained from summing the scores of all items.
Heart rate | 24 weeks
  Beats per minute
Blood pressure | 24 weeks
  mmHg
Measure of body weight | 24 weeks
  Measurements done at visit - weight in kilograms
Measure of body mass index | 24 weeks
  Measurements done at visit - body mass index as per kg/m^2
Measure of waist circumference and hip circumference | 24 weeks
  Measurements done at visit - circumference in cm
Measure of waist-to-hip ratio | 24 weeks
  Measurements done at visit
Lipid profile, specifically: LDL-cholesterol, HDL-cholesterol, triglycerides | 24 weeks
  Blood tests, in mmol/L
Urine albumin-creatinine ratio | 24 weeks
  Urine test

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (that is, insulin delivery, glucose levels and individual participant data) and informed consent form will be shared by the corresponding author, for academic purposes, subject to a material transfer agreement and approval of the McGill University Health Center's Research Ethics Board. All data shared will be de-identified. Raw data will be shared for non-commercial use upon reasonable request and a material transfer agreement.
Supporting Information: ICF